CLINICAL TRIAL: NCT01881685
Title: Fetal Intrapartum Heart Rate FHR/ECG Study
Status: Completed | Type: Observational
Sponsor: Mindchild Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP#12018
Record Dates: First submitted 2013-06-11; First posted 2013-06-20 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2014-09

CONDITIONS: Abnormality in Fetal Heart Rate or Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — 1) umbilical cord arterial and venous blood; 2)placenta for pathological evaluation.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to evaluate the association between certain markers in the blood of neonatal brain injury and specific Fetal Heart Rate monitoring findings using the device under study.

DETAILED DESCRIPTION:
The purpose of the study is to:

1. evaluate the association between serologic markers of neonatal brain injury and the specific FHR monitoring findings using the investigational device;
2. investigate the relationship between selective serotonin reuptake inhibitor (SSRI) antidepressants and the QT interval of the fetal heart. Specifically, examine the potential association between maternal SSRI use and the fetal QT interval,and;
3. develop the capacity to measure uterine contractions during labor using non-invasive electrodes that measure the electrical signal from the uterine muscle.

For this study, the investigational device will not be used to diagnose or treat as it will be used in concert with the current standard of care monitors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester and Women in labor (the progressive effacement and dilatation of the cervix) who are having their fetus' heart rate monitored continuously will form the eligible population for recruitment into our study
* 18 years old or older
* Women with the diagnosis of fetal intrauterine growth restriction may be included.

Exclusion Criteria:

* Speakers of languages other than English
* Gestational age less than 24 weeks 0 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in labor who are having their fetus' heart rate monitored continuously
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quantitative FHR patterns predictive of adverse neonatal outcome | During Labor
  1)quantitative analysis of fetal heart-rate (FHR) data recorded during labor using advanced mathematical techniques, including pattern-recognition analysis using EKG stickers applied to the maternal abdomen.

SECONDARY OUTCOMES:
Uterine contraction measurement | During Labor
  Uterine contraction monitoring using skin surface electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Drake, MD, Principal Investigator — Summa Center for Women's Health Research
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Summa Center for Women's Health Research, Akron, Ohio